CLINICAL TRIAL: NCT06564051
Title: A Prospective Observational Study to Assess Monoclonal B-Cell Lymphocytosis in Individuals With Chronic Hepatitis C
Brief Title: Study to Assess Monoclonal B-Cell Lymphocytosis in Individuals With Chronic Hepatitis C
Status: Terminated | Type: Observational
Why Stopped: slow accrual
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 17-003975; NCI-2024-01768 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 17-003975 (Other: Mayo Clinic Institutional Review Board)
Record Dates: First submitted 2024-08-19; First posted 2024-08-21 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Chronic Viral Hepatitis C; Monoclonal B-Cell Lymphocytosis
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples retained only with participant permission
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood sample collection and have medical records reviewed throughout study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the incidence of monoclonal B-cell lymphocytosis MBL) in patients with chronic hepatitis C and to determine if monoclonal b-cell lymphocytosis is affected by treatment for hepatitis C.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the prevalence of MBL in patients with chronic hepatitis C who are to begin therapy with directly acting antiviral (DAA), and compare with clinic controls who are seen in the general medicine clinic at Mayo Clinic.

II. To determine the correlation between the specific subtype of MBL (CD5- MBL, atypical CLL-phenotype MBL and CLL-phenotype MBL) relative to the hepatitis C virus (HCV) genotype.

III. To assess the proportion of individuals with MBL who have an improvement in the circulating monoclonal B-cell population following therapy with DAA.

OUTLINE: This is an observational study.

Patients undergo blood sample collection and have medical records reviewed throughout study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with chronic hepatitis C who are to begin therapy with DAA

  * Willing to submit a peripheral blood sample at baseline, end of therapy, 12 weeks after the end of therapy, and 52 weeks from baseline

Exclusion Criteria:

* Individuals with chronic hepatitis C who have cirrhosis

  * Individuals with chronic hepatitis C who have a past history of a lymphoproliferative disorder AND for which they received chemotherapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with hepatitis C who are to begin therapy with DAA seen in the Division of Gastroenterology and Hepatology at Mayo Clinic in Rochester.
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2025-12-03 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Prevalence of monoclonal B-cell lymphocytosis (MBL) | Baseline; up to one year
  Blood samples collected in conjunction with routine clinical blood draws will be tested for MBL and compared with post-therapy samples and with control patients (without hepatitis C).

CONTACTS AND LOCATIONS:
Overall Officials: Sameer A. Parikh, M.B.B.S., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials